CLINICAL TRIAL: NCT06388629
Title: Epicardial Access Study With Rook (EASY-R)
Brief Title: Epicardial Access Study With Rook
Acronym: EASY-R
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Circa Scientific, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M064-066 Rev 00
Record Dates: First submitted 2024-04-20; First posted 2024-04-29 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Arrythmia
Keywords: Electrophysiology; Pericardial Access; Epicardial Access; EP
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Experimental): Single arm of the study that receives treatment with the subject device.
  Interventions: Device: Rook Epicardial Access Kit

INTERVENTIONS:
Device: Rook Epicardial Access Kit — Access the epicardial surface of the heart via a subxiphoid approach with the subject device to facilitate guidewire placement into the pericardium.

SUMMARY:
The goal of this clinical trial is to test how how effective the Circa Scientific Rook® Epicardial Access Kit is at gaining guidewire access to the outside surface of the heart (epicardium). In addition the safety of the device will be compared to the available data for alternative methods of epicardial access.

Participants will receive treatment with the subject device during the course of a typical epicardial electrophysiology procedure.

DETAILED DESCRIPTION:
This trial is a confirmatory trial for the Circa Scientific Rook® Epicardial Access Kit for accessing the epicardial surface of the heart via a subxiphoid approach to facilitate guidewire placement into the pericardial space in adult patients. The purpose of this study is to confirm the safety and establish the efficacy of the Circa Scientific Rook® Epicardial Access Kit as a pericardial access device. The Rook® Epicardial Access Kit will be used to gain access the epicardial surface of the heart via a subxiphoid approach in adult patients with a normal, non-distended pericardial space.

Access success of the test device to the pericardial space and occurrence of CEC-adjudicated device and procedure related adverse events will be assessed in relation to complication rate existing data from the literature presenting epicardial access procedure results during subxiphoid (minimally invasive) surgical procedures. This is a prospective, single-arm, non-randomized study.

The primary endpoint is successful pericardial access through the use of the Circa Scientific Rook® Epicardial Access Kit, achieving guidewire access to the pericardial space as confirmed during the procedure by standard x-ray technique. The safety endpoint is the occurrence of CEC-adjudicated device or procedure related adverse events through hospital discharge or up to 4 days post procedure, whichever comes first. Additional endpoints include speed of access, ease of use and human factors data.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is clinically indicated to undergo a procedure that requires percutaneous access to the normal, non-distended, pericardial space.
2. Patient is willing and able to provide written informed consent.

Exclusion Criteria:

1. Subject is younger than 18 years of age
2. Previous cardiac surgery
3. Myocardial infarction within 4 weeks prior to procedure
4. Class IV NYHA (New York Heart Association) heart failure symptoms
5. Subject with an active systemic infection
6. Known carotid artery stenosis greater than 80%
7. Presence of thrombus in the left atrium
8. Congenital absence of a pericardium
9. Coagulopathy
10. Hemodynamic Instability
11. Acute conditions (i.e. electrolyte abnormality, acute ischemia, drug toxicity)
12. Severe hepatic dysfunction or enlargement
13. Subject has Body Mass Index > 40
14. Life expectancy less than 6 months
15. Subject is pregnant
16. Subject is currently participating in another investigational drug or device study that clinically interferes with the endpoints of this study
17. Subject has known or suspected allergy to contrast media
18. Subject is known to have pericardial fibrosis, pericardial adhesions, or prior failed epicardial access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-17 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Successful Epicardial Access | During procedure.
  The number and percentage of patients in which successful epicardial access is achieved

SECONDARY OUTCOMES:
Speed of Access | During procedure.
  The time from skin incision to confirmed guidewire access to the pericardial space
Rate of Use Errors | During procedure.
  Recording any use errors that may occur in the clinical environment that have not been otherwise been observed.

OTHER OUTCOMES:
Rate of Adverse Events | Patients are monitored for adverse events until hospital discharge or up to 4 day after procedure.
  The rate of occurrence of adverse events that have been determined to be related to the device by the clinical events committee

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, MD, Principal Investigator — Nemocnice Na Homolce
Locations (1):
- Na Homolce Hospital, Prague, Czechia